CLINICAL TRIAL: NCT02150174
Title: Retrieval Practice in Patients With Schizophrenia : an Exploratory Study Using Word Pairs
Brief Title: Testing Effect and Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5806
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia; Episodic Memory Deficits
Keywords: Schizophrenia; Episodic memory deficits
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with schizophrenia (Experimental)
  Interventions: Behavioral: Retrieval practice effect using word pairs and cued recall tests with feedback
- Healthy subjects (Active Comparator)
  Interventions: Behavioral: Retrieval practice effect using word pairs and cued recall tests with feedback

INTERVENTIONS:
Behavioral: Retrieval practice effect using word pairs and cued recall tests with feedback — In the first phase (encoding), people study a list of 48 word pairs non semantically associated.
  Then (initial test), they recall half of word pairs or restudy the other half.
  In the second phase (final test) which takes place 2 days later, they recall all the 48 the word pairs.

SUMMARY:
When people are tested on a previously learned material, they will latter remember it better even when compared to a condition where they can re-study it. This phenomenon is called retrieval practice and is supported by an extensive research literature mostly carried out in normal students. This paradigm begins to be used in cognitive remediation programs in patients suffering from memory difficulties.

The objective of this study is to investigate whether retrieval practice is spared in patients with schizophrenia.

If effective, this method could be used in cognitive remediation programs.

Since episodic memory difficulties are supposed to be secondary to deficits in the initiation/elaboration of efficient encoding and retrieval strategies our hypothesis is that retrieval practice is spared in schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* French is the native language, or acquired before 5 years old
* People must be able to understand and follow the trial instructions

Specific inclusion criteria (for patients) :

* Diagnostic of schizophrenia, according to the DSM -5, clinically stable
* The treatment must remain unchanged during the trial

Exclusion Criteria:

* Severe or acute cerebral disease
* Other actual psychiatric disorder
* Use of drugs with high anticholinergic effect
* Irregular use of benzodiazepines medication, or high dose of benzodiazepin (more than 2 mg of lorazepam per day or equivalent)
* Inappropriate use of drugs

Specific exclusion criteria (for healthy subjects) :

- Diagnostic of schizophrenia of a relative up to the third degree

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of word pairs properly recalled | Final test : 2 days after the first experimental session
  - The aim is to investigate the retrieval practice effect using word pairs and cued recall tests with feedback in patients with schizophrenia and healthy controls.
  In the first phase (encoding), people study a list of 48 word pairs non semantically associated, then half of the pairs are presented in its completed form for two times, and for the other half the two subsequent re-exposure trials are framed as cued recall tests (the first word is presented and the subject has to remember and give orally the second word, and a feedback is given).
  In the second phase (final test) which takes place 2 days later, all the 48 word pairs are presented as a cued recall test.
  - We will compare in patients with schizophrenia and healthy controls final performance recall for information studied and recalled ("test" condition) to those for information studied and then re-studied ("re-study" condition).

SECONDARY OUTCOMES:
Difference between final performance recall and memory span score | Final test : 2 days after the first experimental session
  In each group (patients with schizophrenia and healthy controls) :
  Difference between the final performance recall (see primary outcome measure) in "test" condition and "re-study" condition AND memory span score.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Psychothérapique de Nancy, Laxou
  - Service de psychiatrie - Hôpital Civil - CHRU Strasbourg, Strasbourg

REFERENCES:
- [Result] Jantzi C, Mengin AC, Serfaty D, Bacon E, Elowe J, Severac F, Meyer N, Berna F, Vidailhet P. Retrieval practice improves memory in patients with schizophrenia: new perspectives for cognitive remediation. BMC Psychiatry. 2019 Nov 11;19(1):355. doi: 10.1186/s12888-019-2341-y. PMID 31711448